CLINICAL TRIAL: NCT06719934
Title: Dienogest Versus Uterine Artery Embolization in Ttt of Adenomyosis -cohort Comparetive Study
Brief Title: Ttt of Adenomyosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Eshraq Arabi, Assuit, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121212121212121212121212121212
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — dienogest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dienogest group (Experimental): will take 2 mg oral Dienogest
  Interventions: Drug: Dienogest 2 mg orally
- Uterine artery embolization (Experimental): will undergoes uterine artery embolization by local anasthesia
  Interventions: Procedure: UAE

INTERVENTIONS:
Drug: Dienogest 2 mg orally — 2 mg Dienogest orally
  Arms: Dienogest group
Procedure: UAE — under local anasthesia uterine artery embolizationwill be done
  Arms: Uterine artery embolization

SUMMARY:
to evaluate use of Dienogest versus uterine arteries embolization in treatment of Adenomyosis-associated symptoms as dysmenorrhea, heavy menstrual bleeding and bulk-related symptoms

DETAILED DESCRIPTION:
Type of the study: prospective cohort comparative study. Setting: It will be done at both Obstetrics & Gynecology department and Radiology department, Al-Azhar University Hospital Assiut branch.

Time of the study: Starting from January 2025 till the end of the study Number of cases: 100 cases. According to sample size equation Where; in: n = number of patients, = 1.96 (standard normal deviate value that divides the central 95% of z distribution from 5% in the tails), P = the reported sensitivity (67%, i.e., 0.67), L= absolute precision desired on either side (half width of the confidence interval of the confidence interval) of sensitivity (10% i.e., 0.1).

Inclusion criteria:

* Age Group: 30-50 years
* Women with adenomyosis
* With or without small fibroids
* Suffering from heavy menstrual bleeding, dysmenorrhea, and/or cycle- independent pain and bulk-related symptoms.

Exclusion criteria:

* Presence of a malignancy or pelvic infection.
* An on-going pregnancy or a desire to conceive in the future.
* Absolute contraindication for angiography (renal impairment).
* Chronic debilitating diseases.

ELIGIBILITY:
Inclusion Criteria:- Age Group: 30-50 years

* Women with adenomyosis
* With or without small fibroids
* Suffering from heavy menstrual bleeding, dysmenorrhea, and/or cycle- independent pain and bulk-related symptoms.

Exclusion Criteria:

* - Presence of a malignancy or pelvic infection.
* An on-going pregnancy or a desire to conceive in the future.
* Absolute contraindication for angiography (renal impairment).
* Chronic debilitating diseases.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
evaluation use of Dienogest versus uterine arteries embolization in treatment of Adenomyosis-associated symptoms as dysmenorrhea, heavy menstrual bleeding and bulk-related symptoms by questionnaire | through study completion ,an average of 1 year
  evaluation use of Dienogest versus uterine arteries embolization in improvement of Adenomyosis-associated symptoms as dysmenorrhea, heavy menstrual bleeding and bulk-related symptoms by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No